CLINICAL TRIAL: NCT07350330
Title: Comparative Study of Muscle Transplantation Versus Y Splitting Recession Technique in Treatment of Large Angle Exotropia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD223/2025
Record Dates: First submitted 2025-12-20; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Exotropia
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle transplantation (Active Comparator): This group will undergo medial rectus resection, lateral rectus recession, with muscle transplantation
  Interventions: Procedure: muscle transplantation
- Y splitting (Active Comparator): This group will undergo medial rectus resection, lateral rectus recession, with Y splitting
  Interventions: Procedure: Y splitting

INTERVENTIONS:
Procedure: muscle transplantation — transplanting a resected part of medial rectus to the already recessed lateral rectus muscle
  Arms: Muscle transplantation
Procedure: Y splitting — Y splitting of the recessed lateral rectus muscle
  Arms: Y splitting

SUMMARY:
This study is designed to correct large-angle exotropia by monocular surgery. It compares two augmented recession techniques, which are recession with muscle transplantation and recession with Y splitting.

ELIGIBILITY:
Inclusion Criteria:

* Age should be of more than 6 years Exotropia of an angle ranging from 50 to 70 PD Myopic or hypermetropic refraction

Exclusion Criteria:

* history of previous squint surgery significant vertical deviation incomitant squint in the form of paralytic or restrictive disorder any neurological disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Ocular alignment | from the operation till six months postoperatively
  To measure ocular alignment using prisms after lateral rectus recession with muscle transplantation versus lateral rectus recession with Y splitting

SECONDARY OUTCOMES:
palpebral fissure height | from preoperative to 6 months postoperative
  Assess whether this is a change in palpebral fissure height pre- and postoperatively by measurement using a ruler
ocular incomitance | from surgery till 6 months afterward
  The presence of ocular incomitance and gaze restriction using prisms and motility tests after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided